CLINICAL TRIAL: NCT04997187
Title: Effect of Bacillus Coagulans on Various Symptoms and Fecal Microbial Diversity in Adults With With Functional Constipation: a Randomized, Double-blinded, Placebo-controlled Trial
Brief Title: Effect of Bacillus Coagulans in Adults With With Functional Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Sang Yeoup Lee, Professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 02-2021-008
Record Dates: First submitted 2021-07-30; First posted 2021-08-09 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2023-04

CONDITIONS: Constipation - Functional
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bacillus coagulans group (Experimental): This group takes Bacillus coagulans for 12 weeks.
  Interventions: Dietary Supplement: Bacillus coagulans group
- Control group (Placebo Comparator): This group takes placebo for 12 weeks.
  Interventions: Dietary Supplement: Control group

INTERVENTIONS:
Dietary Supplement: Bacillus coagulans group — Bacillus coagulans 400 mg/day for 12 weeks
  Arms: Bacillus coagulans group
Dietary Supplement: Control group — Placebo 400 mg/day for 12 weeks
  Arms: Control group

SUMMARY:
The investigators conduct a randomized, double-blind, placebo-controlled study to investigate the effects of Bacillus coagulans on various symptoms and fecal microbial diversity in adults with with functional constipation for 12 weeks.

DETAILED DESCRIPTION:
A previous study has indicated that Bacillus coagulans provided control of abdominal pain, less discomfort during defecation, and a more normalized defecation style, especially in adults with with functional constipation. Therefore, the investigators conduct a randomized, double-blind, placebo-controlled study to investigate the effects of Bacillus coagulans various symptoms and fecal microbial diversity in adults with with functional constipation for 8 weeks; the safety of the compound are also evaluated. The Investigators examine constipation visual analogue scale, Bristol Stool Form Scale type 3 & 4 ratio, visual analogue scale for irritable bowel syndrome (VAS-IBS) questionnaire score, IBS-symptom severity scale, IBS quality-of-life questionnaire score, fecal microbial diversity at baseline, as well as after 8 weeks of intervention. Eighty adults were administered either 400 mg of Bacillus coagulans or a placebo each day for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

- function constipation by Romes criteria IV

Exclusion Criteria:

* Abnormal liver or renal function (more than twice the normal upper limit of the research institute)
* Uncontrolled diabetes mellitus (>160 mg/dL of fasting blood sugar)
* Uncontrolled hypertension (>160/100 mmHg)
* Uncontrolled thyroid diseases.
* History of serious cerebro-cardiovascular diseases or cancer such as angina or myocardial infarction within 6 months
* History of structural abnormalities of colon within 4 year
* History of medication for probiotics and psychiatric diseases such as severe depression, schizophrenia, drug intoxication.
* Alcohol abuser
* Allergic reaction to this test food
* Those who participated in other drug clinical trials within 1 month from the screening date.
* Severe gastrointestinal symptoms such as heartburn and indigestion
* Those who are pregnant, lactating, or plan to become pregnant during the clinical trial
* Those who are judged to be unsuitable by the PI for other reasons

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2022-02-27 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
constipation visual analogue scale | 8 weeks
  using visual analogue scale (100 mm). The minimum value was 0 mm and the maximum value was 100 mm, and higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Bristol Stool Form Scale (BSFS) type 1 & 2 ratio (%) | 8 weeks
  using Bristol Stool Form Scale. The minimum value was 0% and the maximum value was 100%, and higher scores mean a better outcome.
visual analogue scale for irritable bowel syndrome | 8 weeks
  using visual analogue scale (100 mm). The minimum value was 0 mm and the maximum value was 100 mm, and higher scores mean a better outcome.
irritable bowel syndrome-symptom severity scale | 8 weeks
  using IBS-Symptom Severity Scale questionnaire. The minimum value was 0 score and the maximum value was 500 score and higher scores mean a worse outcome.
irritable bowel syndrome-quality-of-life | 8 weeks
  using IBS-QOL questionnaire. The minimum value was 0 score and the maximum value was 5 score and higher scores mean a better outcome.
fecal microbial diversity | 8 weeks
  using gut microbiome analysis

CONTACTS AND LOCATIONS:
Overall Officials: Sang Yeoup Lee, MD, PhD, Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, Gyeungsangnam-do, South Korea

IPD SHARING:
Plan to Share IPD: No